CLINICAL TRIAL: NCT03203252
Title: Pilot Study Towards Development of an Objective Evaluation of Outcome After Implant-based Breast Reconstruction, Using 3D-surface Imaging (3D-SI) and the Feasibility of a Novel Online Research Tool.
Brief Title: Pilot Study for 3-Dimensional Surface Imaging in Implant-based Breast Reconstruction
Acronym: 3D-SI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4707
Record Dates: First submitted 2017-06-15; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reconstruction BREAST-Q — Validated Patient reported outcome measure specifically designed to assess Quality of life domains and satisfaction following breast reconstruction.
Other: 3-dimensional Surface Image — Non-invasive 3-dimensional photograph using VECTRA® XT 3D imaging system.
Other: Treatment Questionnaire — Online questionnaire pertaining to treatment received pertaining to breast cancer or risk reduction for breast cancer.

SUMMARY:
Measuring appearance of implant-based breast reconstruction after mastectomy for breast cancer - an online approach to research. Using 3-dimensional surface images we intend to create a tool to measure appearance after surgery in order to improve standards of care for women. We want to minimise the number of visits and amount of time involved in research participation so this pilot study will develop new online tools for information giving and gathering, and for consent so that only one visit to hospital will be required for photographs. This will also extend the availability of expensive 3D technology to more women.

DETAILED DESCRIPTION:
Aim To test the feasibility of a number of novel initiatives prior to their use in a multi-centre study. The future study will develop a way to measure cosmetic outcome for implant-based breast reconstruction using 3-dimensional Surface Imaging (3D-SI).

Methods At The Royal Marsden Hospital in Sutton 125 implant-based reconstructions are performed per year (data from 2014). The study team would like to invite women who have had their treatment within the previous 1-5 years to participate in the pilot. The women can be identified through operation records. The study team will aim to include 50.

A letter of invitation will be sent by post. This will include a participant information leaflet, a link to the website, and a unique study ID for each participant. In recent studies, more than 8 out of ten women who were asked to participate agreed.

The website will have the following features:

* Patient study information including links to other relevant information sources (e.g. ABS, Breast Cancer Care, RMH, ICR, BRC), patient testimonials, and biographies from the study team.
* An online consent process for the study.
* A questionnaire for patient demographics (height, weight etc)and treatment information (i.e. type of operation and other treatments like radiotherapy).
* An online version of the BREAST-Q reconstruction module and radiotherapy module from the breast conserving surgery BREAST-Q (a questionnaire designed to assess quality of life and satisfaction with care for patients having breast surgery).
* An online calendar to book a 3D-SI appointment at the hospital.
* A user survey to gain patient feedback on the website and the concept of online consent.
* A 'contact us' section in case further information is required.

At each stage the participant will enter their unique study ID so all of the information collected will remain anonymous. We will hold the code for study IDs securely. There is no patient identifiable data collected on the website. The participant will be guided through the different aspects of the online recruitment processes outlined above. When they have read the patient information, they can click on the link to consent to the study at which point a check screen will ask:

1. I have had enough information and wish to consent to the study - link to the consent form
2. I would like further information which is not available on the website - link to contact us section

Only then will they be able to access the data collection stages of the website and book a photography slot, thereby we can be sure that no patient starts to enter information or attends for a photograph without valid consent.

Following this the participant will be required to attend the hospital only once for an appointment (booked online) for a 3D photograph and height and weight measurement. This will take less than 20 minutes. This will be the end of the patient involvement in the study.

Success in this pilot will provide:

* A bespoke website to facilitate online patient education, consent, and data collection to streamline research processes.
* Information on uptake rate and specific evaluation of the acceptability of the web system and accuracy of patient entered data.
* Data on the accuracy of the VECTRA software to measure implant base reconstruction.
* A secure online 3D-SI storage facility to enable access from multiple hospitals to enable wider involvement in large scale research.
* A library of 3D-surface images on which to base a panel assessment score for implant-based reconstruction by way of a consensus meeting at the outset of the future multi-centre study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Over 18 years
* Have undergone implant-based reconstruction 1-5 years before study entry (can be unilateral or bilateral, immediate or delayed, nipple-sparing or nipple-sacrificing, risk reducing or therapeutic)

Exclusion Criteria:

* <1 year or over 5 years from surgery
* Explantation
* Local or distant recurrence
* Lacks capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of female participants who have undergone mastectomy and implant-based reconstruction within the last 1-5 years. The research will be carried out at the Royal Marsden NHS Foundation Trust Sutton.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate to a study of this design | 3 months
  The study team will assess the number of participants as a proportion of those approached. The study team will assess the proportion of those approached versus those who complete the recruitment process by attending for their 3D-SI.

SECONDARY OUTCOMES:
To understand dropout rates | 6 months
  Dropout rate - participants who complete the online recruitment process as a proportion of the number who start the process i.e. those who consent to the study versus those who progress through to booking their photography slot. The user survey is not a compulsory part of the study, therefore if it is not filled it will not preclude women from completing the study by having a 3D-SI.
To understand how long it takes to complete the online recruitment process. | 6 months
  Time taken to complete the entire online process from first log on to completion of evaluation survey.
To understand reasons for not completing the online process once started. | 6 months
  Qualitative information on reasons for not completing once started.
To analyse how accurately participants report data pertaining to their medical treatment and themselves (eg height and weight/use of radiotherapy) | 6 months
  Accuracy of reporting e.g. for yes/ no questions such as 'Did you have radiotherapy after breast reconstruction?' will be represented as the percentage of correct answers (should be >95%).
  For continuous data e.g. weight we will assess the proportion of answers within 5kg of correct answer and for height, the proportion within 5cm/2 inches. This will be represented as a dichotomous within/not within range for analysis, but a range of accuracy will also be reported.
To assess inter- and intra-observer variability in a range of objective measurements to enable us to choose those to measure in the multi-centre study. | 6 months
  For which objective measurements are the inter- and intra-observer variation within 10% Based on previous findings this is an acceptable level of variation. Measures with a greater variation will not be useful in a multi-centre study with more observers and should therefore be avoided.
To assess the feasibility of an online secure storage facility for 3D surface images i.e. how long it takes to upload and evaluate the images, how user-friendly is it? | 6 months
  Time taken to upload and analyse 10 images for a single observer. In one sitting the observer will log onto the program, upload, and analyse each image once (as would be done in the panel assessment). The time will start from the logon and finish when the observer logs out at the end of the 10th image analysis. The mean time taken will be reported. Qualitative data on user friendliness will be gathered to inform improvements in the process by issuing surveys to a test team of medical professionals at the Royal Marsden Hospital with experience in using the VECTRA so the use of the data storage system is the only variable.
To assess the feasibility of online patient satisfaction and quality of life questionnaires. | 6 months
  The BREAST-Q has a pre-and a post-operative section. The post-operative section will be used for this study. The reconstruction module has 14 post-operative domains, each with sub-scales rated 1-4. Domains 7-9 will not be used as these are in reference to autologous reconstruction, domain 10 will only be appropriate for women who have had nipple reconstruction, domains 11-14 are pertaining to satisfaction with information and staff which is not relevant to this study so will not be assessed. The Breast Conserving Therapy Post-operative module domain 2, subscales a-g will be used for women who have undergone radiotherapy. The main point of the exercise in the pilot study will be to ensure the BREAST-Q data can be collected online and analysed. The results will only be for 50 patients so will not be generalisable.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pusic et al. Measuring Quality of Life in Breast Surgery: Content development of a new modular system to capture patient reported outcomes (The MSKCC BREAST-Q). ISOQOL Annual Meeting. October 2006 Lisbon, Portugal
- [Result] Pusic AL, Chen CM, Cano S, Klassen A, McCarthy C, Collins ED, Cordeiro PG. Measuring quality of life in cosmetic and reconstructive breast surgery: a systematic review of patient-reported outcomes instruments. Plast Reconstr Surg. 2007 Sep 15;120(4):823-837. doi: 10.1097/01.prs.0000278162.82906.81. PMID 17805107
- [Derived] Godden AR, Wood SH, James SE, MacNeill FA, Rusby JE. A scoring system for 3D surface images of breast reconstruction developed using the Delphi consensus process. Eur J Surg Oncol. 2020 Sep;46(9):1580-1587. doi: 10.1016/j.ejso.2020.05.016. Epub 2020 Jun 7. PMID 32620404
- See also: BREAST-Q Information — https://eprovide.mapi-trust.org/instruments/breast-q